CLINICAL TRIAL: NCT03027557
Title: Treatment of Primary Hyperparathyroidism With Denosumab and Cinacalcet.
Acronym: DENOCINA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Peter Vestergaard (Other)
Collaborators: Aalborg University (Other)
Responsible Party: Sponsor-Investigator, Peter Vestergaard, Professor, DMSc, Consultant, Aalborg University Hospital
Organization: Aalborg University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 180987; 2016-001510-20 (EudraCT Number)
Record Dates: First submitted 2017-01-16; First posted 2017-01-23 (Estimated); Results first posted 2021-05-25 (Actual); Last update posted 2021-05-25 (Actual); Status verified 2021-05

CONDITIONS: Primary Hyperparathyroidism; Parathyroid Adenoma; Parathyroid Hyperplasia
Keywords: Primary Hyperparathyroidism; Parathyroid Adenoma; Parathyroid Hyperplasia; Cinacalcet; Denosumab; Drug Therapy; Bone Mineral Density; Calcium
MeSH Terms: conditions — Hyperparathyroidism, Primary; Parathyroid Neoplasms | interventions — Cinacalcet; Tablets; Denosumab; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Combined treatment. (Experimental): 20 subjects will be treated with combined 60mg denosumab bi-annually , 30 mg cinacalcet daily and 50 micrograms vitamin-D daily.
  Interventions: Drug: Cinacalcet 30 mg Tablet; Drug: Denosumab Inj 60 mg/ml
- Monotherapy (Active Comparator): 20 subjects will receive 60mg denosumab bi-annually, placebo and 50 micrograms vitamin-D daily.
  Interventions: Drug: Denosumab Inj 60 mg/ml; Other: Placebo tablets
- Placebo (Placebo Comparator): 20 subjects will receive a saline injection bi-annually (blinded), placebo-tablets and 50 micrograms vitamin-D daily.
  Interventions: Other: Placebo tablets; Other: Saline Injection (Placebo)

INTERVENTIONS:
Drug: Cinacalcet 30 mg Tablet — Participants in one arm will receive 30 mg cinacalcet each day.
  Other Names: Mimpara; Sensipar
  Arms: Combined treatment.
Drug: Denosumab Inj 60 mg/ml — Participants in two arms will receive 60 mg Denosumab biannually.
  Other Names: Prolia; Xgeva
  Arms: Combined treatment.; Monotherapy
Other: Placebo tablets — Participants in two arms will receive one placebo-tablet each day.
  Arms: Monotherapy; Placebo
Other: Saline Injection (Placebo) — Participants in one arm will receive saline injections as placebo for denosumab.
  Other Names: Sodium Chloride (NaCl) Fresenius "Kabi"
  Arms: Placebo

SUMMARY:
The only known cure for primary hyperparathyroidism is surgical removal of one or more parathyroid glands. Some patients however, do not fulfill criteria for surgery or do not want to undergo a procedure due to fear of the associated risks. Therefore a medical alternative is warranted.

This study aims to evaluate the effects of Denosumab alone, and in combination with Cinacalcet, as a medical treatment for patients suffering from primary hyperparathyroidism, with mild osteoporosis. To the best of our knowledge no previously reported randomized controlled trial has investigated the use of denosumab in primary hyperparathyroidism.

60 patients will be enrolled in three different treatment-groups: 20 receiving both Denosumab and Cinacalcet, 20 Denosumab and placebo and 20 placebo and placebo. Patients included do not meet the criteria for, or have no wish for a surgical procedure.

By combining the two drugs, this study could possibly contribute to the discovery of a realistic medical alternative to surgery. It is expected that the therapy will be able to both control s-calcium and s-intact parathyroid hormone (iPTH), and simultaneously enhance bone-structure. The therapy thus has the potential of preventing fractures and possibly other long-term effects of primary hyperparathyroidism such as formation of kidney stones, and coronary calcification. Another objective of this project is to investigate whether the combined therapy can facilitate an actual reset of the Calcium-sensing receptor, and thereby de facto cure the disease.

DETAILED DESCRIPTION:
Background/Context:

This project deals with medical treatment of primary hyperparathyroidism. The only cure currently available is surgical removal of one or more parathyroid glands, but this option is neither feasible, nor desirable in all patients with the diagnosis.

Today a major group of patients are being diagnosed by coincidence with biochemical blood-screening, and are therefore in an asymptomatic state of the disease at the time of diagnosis. Long term studies show that these patients over time often have progression in their disease, and develop complications such as osteoporosis. Thus a medical alternative is warranted.

Previous studies have investigated the effects of well known antiresorptive drugs such as bisphosphonates, as well as estrogen-related compounds. These drugs have had effects on particularly bone mineral density (BMD) and biochemical bone-turnover markers, but have been able only transiently to lower blood-calcium levels. Combined with too many unwanted side-effects and a high prevalence of contraindications for a large proportion of the patients needing treatment, these drugs have not provided a realistic alternative to surgery.

Treatment today generally follows the international consensus for treatment of asymptomatic patients with primary hyperparathyroidism. Briefly this includes watchful waiting with biannual control-sessions for indication of surgery, screening for kidney stones/nephrolithiasis, osteoporosis and s-calcium - and s-iPTH levels.

This randomized controlled trial involves the drugs Cinacalcet og Denosumab. Denosumab has previously been shown to greatly improve BMD, lower s-calcium, lower the rate of bone-turnover and prevent osteoporotic fractures in several populations with different diseases, but has never been tested in a published randomized controlled trial in patients with primary hyperparathyroidism.

Cinacalcet has been proved able to lower s-iPTH, lower s-Calcium and thereby relieve symptoms of hypercalcaemia caused by primary hyperparathyroidism. It does not however, lower the rate of bone turnover, and it has not been show to improve BMD.

By combining the two drugs, this study could possibly contribute to the discovery of a realistic medical alternative to surgery. It is expected that the therapy will be able to both control s-calcium and s-iPTH, and simultaneously enhance bone-structure. The therapy thus has the potential of preventing fractures and possibly other long-term effects of primary hyperparathyroidism such as formation of kidney stones, and coronary calcification. Another objective of this project is to investigate whether the combined therapy can facilitate an actual reset of the Calcium-sensing receptor, and thereby de facto cure the disease.

ELIGIBILITY:
Inclusion Criteria:

* Men and women of 18 years of age or older.
* T-score by Dual X-ray Absorptiometry (DXA) between -1,0 og -3,5
* Patients from The North Jutland Region diagnosed with primary hyperparathyroidism at the Department of Endocrinology, Aalborg University Hospital. (Hypercalcaemia measured at two different time-points and simultaneous elevated/inappropriately high PTH, and exclusion of differential diagnosis.)

Exclusion Criteria:

* Medical history of diseases leading to hypercalcaemia other than Primary Hyperparathyroidism.
* Patients being treated with Denosumab or Cinacalcet prior to inclusion or previously treated with Denosumab or Cinacalcet.
* Moderately - Severely decreased liver function (alanine aminotransferase >250u/l, gamma-glutamyl transferase>150u/l, Bilirubin >30)
* Acute myocardial infarction or apoplexia in the 3 months before inclusion.
* Medical record of heart failure
* Risk factors of prolonged corrected QT interval (QTc).
* Open lesions from oral surgery.
* Primary diseases of the bone other than osteoporosis.
* Patients suffering from kidney disease or renal failure.
* Patients under treatment with thiazide or lithium.
* Medical record of generalized seizures or epilepsy.
* Active malignant disease.
* Known allergies towards the specified medicinal products (IMPs).
* Pregnancy or breastfeeding.
* Fertile women who do not agree to the usage of effective contraception.
* Other circumstances, evaluated by the responsible investigator, making the subject unsuitable for participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-09-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julius Simoni Leere, MD, Principal Investigator — Aalborg University and Aalborg University Hospital; Peter Vestergaard, DMSc, Study Director — Aalborg University and Aalborg University Hospital
Locations (1):
- Aalborg University Hospital, Aalborg, Denmark

REFERENCES:
- [Derived] Leere JS, Karmisholt J, Robaczyk M, Lykkeboe S, Handberg A, Steinkohl E, Brondum Frokjaer J, Vestergaard P. Denosumab and cinacalcet for primary hyperparathyroidism (DENOCINA): a randomised, double-blind, placebo-controlled, phase 3 trial. Lancet Diabetes Endocrinol. 2020 May;8(5):407-417. doi: 10.1016/S2213-8587(20)30063-2. PMID 32333877

RESULTS

PARTICIPANT FLOW:
Groups:
- Combined Treatment.: 15 subjects were treated with combined 60mg denosumab every six months, 30 mg cinacalcet daily and 50 micrograms vitamin-D3 daily.
- Denosumab Monotherapy: 16 subjects received 60 mg denosumab every six months, placebo and 50 micrograms vitamin-D daily.
- Placebo: 15 subjects will receive a saline injection every six months(blinded), placebo-tablets and 50 micrograms vitamin-D daily.
Period: Overall Study
Arm/Group | Combined Treatment. | Denosumab Monotherapy | Placebo
Started | 15 | 16 | 15
Completed | 14 | 16 | 15
Not Completed | 1 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Combined Treatment. | Denosumab Monotherapy | Placebo | Total
Number analyzed (Participants) | 15 | 16 | 15 | 46
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.1 (13.2) | 65.4 (8.8) | 68.0 (7.0) | 66.15 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 13 | 12 | 39
  Male | 1 | 3 | 3 | 7
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Denmark | 15 | 16 | 15 | 46
T-score Lumbar Spine (LS) by Dual X-ray Absorptiometry (DXA) [Mean (Standard Deviation); unit: T-score] — Baseline Bone mineral density (BMD) at lumbar spine (L2-L4) T-score. The T-score is the number of units that the bone density is above or below the average. -1 and above-bone density is considered normal; Between -1 and -2.5-is a sign of osteopenia, a condition in which bone density is below normal and may lead to osteoporosis. -2.5 and below-indicates osteoporosis
  T-score | -1.9 (0.93) | -2.0 (0.68) | -1.3 (0.85) | -1.7 (0.87)
T-score TH (by DXA) [Mean (Standard Deviation); unit: T-score] — Baseline Bone mineral density (BMD) at Total Hip (TH) T-score. The T-score is the number of units that the bone density is above or below the average. -1 and above-bone density is considered normal; Between -1 and -2.5-is a sign of osteopenia, a condition in which bone density is below normal and may lead to osteoporosis. -2.5 and below-indicates osteoporosis.
  T-score | -1.4 (0.5) | -1.4 (0.6) | -1.1 (0.5) | -1.3 (0.5)
T-score FN (by DXA) [Mean (Standard Deviation); unit: T-score] — Baseline Bone mineral density (BMD) at Femoral Neck (FN) T-score. The T-score is the number of units that the bone density is above or below the average. -1 and above-bone density is considered normal; Between -1 and -2.5-is a sign of osteopenia, a condition in which bone density is below normal and may lead to osteoporosis. -2.5 and below-indicates osteoporosis.
  T-score | -2.0 (0.7) | -1.9 (0.7) | -1.7 (0.6) | -1.88 (0.6)
T-score 1/3 FA (by DXA) [Mean (Standard Deviation); unit: T-score] — Baseline Bone mineral density (BMD) at 1/3 distal forearm (1/3 FA)T-score. The T-score is the number of units that the bone density is above or below the average. -1 and above-bone density is considered normal; Between -1 and -2.5-is a sign of osteopenia, a condition in which bone density is below normal and may lead to osteoporosis. -2.5 and below-indicates osteoporosis.
  T-score | -2.4 (1.2) | -2.4 (1.2) | -2.8 (0.9) | -2.5 (1.1)
Volumetric Bone Mineral Density (vBMD) LS [Mean (Standard Deviation); unit: mg/cm^3] — Baseline lumbar spine BMD by quantitative computed tomography (QCT)
  mg/cm^3 | 96.4 (28.1) | 99.7 (24.0) | 94.2 (25.4) | 96.9 (25.1)
vBMD distal forearm [Mean (Standard Deviation); unit: mg/cm^3] — Bone Mineral Density at the distal forearm by QCT
  mg/cm^3 | 183.5 (32.0) | 194.9 (37.6) | 181.4 (35.5) | 192.6 (34.6)
Cortical width [Mean (Standard Deviation); unit: mm] — Baseline cortical Width of the distal forearm.
  mm | 1.23 (0.5) | 1.19 (0.5) | 1.14 (0.4) | 1.2 (0.4)
Nephrolithiasis [Count of Participants; unit: Participants] — Subjects with nephrolithiasis at baseline
  Participants | 0 | 3 | 1 | 4
Nephrocalcinosis [Count of Participants; unit: Participants] — Subjects with nephrocalcinosis at baseline
  Participants | 2 | 1 | 3 | 6
Pancreas calcifications [Count of Participants; unit: Participants] — Subjects with pancreatic calcifications at baseline
  Participants | 0 | 1 | 2 | 3
Fracture by Vertebral Fracture Assessment (VFA) [Count of Participants; unit: Participants] — Subjects with vertebral fractures by VFA at baseline
  Participants | 1 | 3 | 2 | 6
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] — Body Mass Index at baseline
  kg/m^2 | 27.7 (3.5) | 27.4 (4.8) | 28.4 (3.9) | 27.8 (4.0)
Ionized Calcium [Mean (Standard Deviation); unit: mmol/l] — Baseline ionized calcium levels.
  mmol/l | 1.39 (0.08) | 1.39 (0.078) | 1.39 (0.08) | 1.39 (0.06)
P-Parathyroid Hormone (PTH) [Mean (Standard Deviation); unit: pmol/l] — Baseline Parathyroid Hormone level.
  pmol/l | 12.1 (6.2) | 13.1 (6.4) | 11.2 (4.3) | 12.1 (5.7)
Agatston Score [Median (Inter-Quartile Range); unit: units on a scale] — Agatston score is a score based on the extent of coronary artery calcification calculated on the amount of plaque observed in a CT scan. A score of zero indicates absence of coronary calcium, 1-10: minimal calcification, 11-100 mild calcification, 101-400 moderate calcification, >400 severe calcification.
  Thus the score increases with increasing level of calcification in the coronary vessels.
  units on a scale | 4.9 [0.7 to 25.9] | 10.1 [0.3 to 470.3] | 55.7 [6.8 to 144.6] | 15.5 [0.65 to 129.6]
U-Calcium [Median (Inter-Quartile Range); unit: mg/d] — Baseline urine calcium excretion per day.
  mg/d | 338 [159 to 419] | 276 [218 to 555] | 314 [222 to 373] | 284 [218 to 393]
U-Phosphorous [Median (Inter-Quartile Range); unit: mmol/d] — Baseline daily excretion of phosphorous in urine.
  mmol/d | 28.5 [25.7 to 33.6] | 32.2 [26.5 to 37.0] | 35.2 [23.6 to 39.5] | 32.0 [25.6 to 37.9]
P-Phosphorous [Mean (Standard Deviation); unit: mmol/l] — Baseline p-phosphorous.
  mmol/l | 0.77 (0.15) | 0.77 (0.16) | 0.79 (0.12) | 0.78 (0.14)
Major Depression Inventory score [Median (Inter-Quartile Range); unit: MDI-points] — The Major Depression Inventory (MDI) is a mood questionnaire developed by the World Health Organization. To calculate the total score, a sum of ten individual items (each with an individual score between 0-5, with 0 indicating absence of a symptom and 5 indicating constant presence of a given symptom) is used. A higher score signifies deeper depression with 50 being the maximum score.
  MDI-points | 5 [2 to 11] | 5 [1.5 to 8.5] | 5 [2 to 7] | 5 [2 to 8]

OUTCOME MEASURES:

1. Primary Outcome: Change in Lumbar Spine Bone Mineral Density
Description: Change of Bone Mineral Density after one year of treatment from baseline. Measured with Dual-energy X-ray absorptiometry (DXA)-scan.
Time Frame: Baseline,one year
Population: One participant from the combined treatment-group was not included in the analysis due to withdrawal before the final scan.
Measure: Mean (Standard Error); unit: g/cm^2
Arm/Group | Combined Treatment. | Denosumab Monotherapy | Placebo
Number analyzed (Participants) | 14 | 16 | 15
g/cm^2 | 0.030 (0.009) | 0.042 (0.009) | -0.016 (0.007)
Statistical Analysis 1: Comparison: Combined Treatment. vs Denosumab Monotherapy vs Placebo; Test type: Superiority; p < 0.00001, ANOVA

2. Primary Outcome: Change in Total Hip Bone Mineral Density
Description: as for outcome 1
Time Frame: Baseline,one year
Population: One participant from the combined treatment-group was not included in the analysis due to withdrawal before the final scan. One participant from the placebo group did not provide results for this analysis as he/she had had a hip-replacement performed.
Measure: Mean (Standard Error); unit: g/cm^2
Arm/Group | Combined Treatment. | Denosumab Monotherapy | Placebo
Number analyzed (Participants) | 14 | 16 | 14
g/cm^2 | 0.027 (0.006) | 0.021 (0.003) | -0.013 (0.006)
Statistical Analysis 1: Comparison: Combined Treatment. vs Denosumab Monotherapy vs Placebo; Test type: Superiority; p < 0.00001, ANOVA

3. Primary Outcome: Change in Femoral Neck Bone Mineral Density
Description: as for outcome 1
Time Frame: Baseline,one year
Population: as for outcome 2
Measure: Mean (Standard Error); unit: g/cm^2
Arm/Group | Combined Treatment. | Denosumab Monotherapy | Placebo
Number analyzed (Participants) | 14 | 16 | 14
g/cm^2 | 0.023 (0.006) | 0.020 (0.005) | -0.007 (0.006)
Statistical Analysis 1: Comparison: Combined Treatment. vs Denosumab Monotherapy vs Placebo; Test type: Superiority; p = 0.0019, ANOVA

4. Primary Outcome: Change in 1/3 Forearm Bone Mineral Density
Description: as for outcome 1
Time Frame: Baseline,one year
Population: One participant from the combined treatment-group was not included in the analysis due to withdrawal before the final scan. One participant from the denosumab group did not provide results for this analysis as he/she experienced a wrist fracture prior to the final scan.
Measure: Mean (Standard Error); unit: g/cm^2
Arm/Group | Combined Treatment. | Denosumab Monotherapy | Placebo
Number analyzed (Participants) | 14 | 15 | 15
g/cm^2 | 0.005 (0.003) | 0.005 (0.003) | -0.005 (0.004)
Statistical Analysis 1: Comparison: Combined Treatment. vs Denosumab Monotherapy vs Placebo; Test type: Superiority; p = 0.096, ANOVA

5. Primary Outcome: Percentage Change in Lumbar Spine Bone Mineral Density
Description: Percentage change of Bone Mineral Density after one year of treatment from baseline.
  Measured with Dual-energy X-ray absorptiometry (DXA)-scan.
Time Frame: Baseline,one year
Population: as for outcome 1
Measure: Mean (Standard Error); unit: % change
Arm/Group | Combined Treatment. | Denosumab Monotherapy | Placebo
Number analyzed (Participants) | 14 | 16 | 15
% change | 3.6 (1.1) | 5.1 (1.1) | -1.8 (0.8)
Statistical Analysis 1: Comparison: Combined Treatment. vs Denosumab Monotherapy vs Placebo; Test type: Superiority; p = 0.0001, ANOVA

6. Primary Outcome: Percentage Change in Total Hip Bone Mineral Density
Description: as for outcome 5
Time Frame: Baseline,one year
Population: as for outcome 2
Measure: Mean (Standard Error); unit: % change
Arm/Group | Combined Treatment. | Denosumab Monotherapy | Placebo
Number analyzed (Participants) | 14 | 16 | 14
% change | 3.45 (0.72) | 2.64 (0.41) | -1.50 (0.72)
Statistical Analysis 1: Comparison: Combined Treatment. vs Denosumab Monotherapy vs Placebo; Test type: Superiority; p < 0.00001, ANOVA

7. Primary Outcome: Percentage Change in Femoral Neck Bone Mineral Density
Description: as for outcome 5
Time Frame: Baseline,one year
Population: as for outcome 2
Measure: Mean (Standard Error); unit: % change
Arm/Group | Combined Treatment. | Denosumab Monotherapy | Placebo
Number analyzed (Participants) | 14 | 16 | 14
% change | 3.70 (0.98) | 3.03 (0.86) | -0.78 (0.9)
Statistical Analysis 1: Comparison: Combined Treatment. vs Denosumab Monotherapy vs Placebo; Test type: Superiority; p = 0.0027, ANOVA

8. Primary Outcome: Percentage Change in 1/3 Forearm Bone Mineral Density
Description: as for outcome 5
Time Frame: Baseline,one year
Population: as for outcome 4
Measure: Mean (Standard Error); unit: % change
Arm/Group | Combined Treatment. | Denosumab Monotherapy | Placebo
Number analyzed (Participants) | 14 | 15 | 15
% change | 0.94 (0.7) | 0.88 (0.5) | -0.91 (0.7)
Statistical Analysis 1: Comparison: Combined Treatment. vs Denosumab Monotherapy vs Placebo; Test type: Superiority; p = 0.081, ANOVA

9. Secondary Outcome: Change in Volumetric BMD for the Lumbar Spine.
Description: Measured at baseline and after one year by QCT.
Time Frame: Baseline, one year
Population: One participant from the combined treatment-group was not included in the analysis due to withdrawal before the final scan. Another scan could not be included due to a technical problems with the image analysis.
Measure: Mean (Standard Error); unit: mg/cm^3
Arm/Group | Combined Treatment. | Denosumab Monotherapy | Placebo
Number analyzed (Participants) | 13 | 16 | 15
mg/cm^3 | 4.93 (2.15) | 5.35 (1.91) | -2.56 (1.6)
Statistical Analysis 1: Comparison: Combined Treatment. vs Denosumab Monotherapy vs Placebo; Test type: Superiority; p = 0.0071, ANOVA

10. Secondary Outcome: Mean P-calcium During Treatment.
Description: Blood samples were acquired once every 4 weeks for safety-purposes.
Time Frame: Monthly up to one year.
Measure: Mean (Standard Error); unit: mmol/l
Units Other Than Participants: p-calcium measurements
Arm/Group | Combined Treatment. | Denosumab Monotherapy | Placebo
Number analyzed (Participants) | 15 | 16 | 15
Number analyzed (p-calcium measurements) | 210 | 240 | 224
mmol/l | 1.28 (0.007) | 1.38 (0.006) | 1.40 (0.004)
Statistical Analysis 1: Comparison: Combined Treatment. vs Denosumab Monotherapy vs Placebo; Test type: Superiority; p = 0.0001, ANOVA

11. Secondary Outcome: Percent Change From Baseline in P-carboxy-terminal Collagen Crosslinks (CTX)
Description: p-CTX, change from baseline at 48 weeks.
Time Frame: Change from baseline at 48 weeks reported.
Population: One participant from the combined treatment-group was not included in the analysis due to withdrawal before the final blood-sampling.
Measure: Median (Inter-Quartile Range); unit: % change
Arm/Group | Combined Treatment. | Denosumab Monotherapy | Placebo
Number analyzed (Participants) | 14 | 16 | 15
% change | -48.7 [-73.2 to -15.8] | -58.2 [-76.7 to -44.3] | 11.8 [1.96 to 40.0]
Statistical Analysis 1: Comparison: Combined Treatment. vs Denosumab Monotherapy vs Placebo; Test type: Superiority; p = 0.0001, Kruskal-Wallis

12. Secondary Outcome: Median Agatstons Score Final
Description: Simultaneously with QCT-measurements coronary calcification was be assessed. Agatston score is a score based on the extent of coronary artery calcification calculated on the amount of plaque observed in a CT scan. A score of zero indicates absence of coronary calcium, 1-10: minimal calcification, 11-100 mild calcification, 101-400 moderate calcification, >400 severe calcification.
  Thus the score increases with increasing level of calcification in the coronary vessels.
Time Frame: Baseline, one year
Population: Some participant from the combined and placebo groups could not be included in the analysis because they had coronary stents.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Combined Treatment. | Denosumab Monotherapy | Placebo
Number analyzed (Participants) | 12 | 16 | 13
score on a scale | 5.0 [0.0 to 78.1] | 24.3 [0.7 to 602.1] | 117.8 [6.8 to 182.6]
Statistical Analysis 1: Comparison: Combined Treatment. vs Denosumab Monotherapy vs Placebo; Test type: Superiority; p = 0.38, Kruskal-Wallis

13. Secondary Outcome: Patients With Nephrolithiasis Final Scan.
Description: Number of subjects w. renal stones at final scan.
Time Frame: Patients with nephrolithiasis at one year reported.
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Combined Treatment. | Denosumab Monotherapy | Placebo
Number analyzed (Participants) | 14 | 16 | 15
Participants | 0 | 3 | 1

14. Secondary Outcome: Patients With Pancreas-calcifications Final Scan.
Description: By QCT.
Time Frame: Patients with pancreas-calcifications at one year reported.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Combined Treatment. | Denosumab Monotherapy | Placebo
Number analyzed (Participants) | 14 | 16 | 15
Participants | 0 | 1 | 2

15. Secondary Outcome: Reset of the Calcium Sensing Receptor?
Description: Measured from effect on s-calcium and PTH weeks after termination of IMP
Time Frame: 2 weeks after termination of medication.
Reporting Status: Not Posted

16. Secondary Outcome: Vertebral Fracture Assessment - Final Scan
Description: Number of participants with vertebral fractures as assessed by VFA at final scan.
Time Frame: Patients with vertebral fractures at one year reported.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Combined Treatment. | Denosumab Monotherapy | Placebo
Number analyzed (Participants) | 14 | 16 | 15
Participants | 1 | 3 | 2

17. Secondary Outcome: Change MDI-score
Description: Major Depression Inventory (MDI)-score, Baseline, 6 months, one year (week 52)., change between baseline and 1 year reported.
  The Major Depression Inventory (MDI) is a mood questionnaire developed by the World Health Organization. To calculate the total score, a sum of ten individual items (each with an individual score between 0-5, with 0 indicating absence of a symptom and 5 indicating constant presence of a given symptom) is used. A higher score signifies deeper depression with 50 being the maximum score.
Time Frame: Baseline, 6 mths, one year.
Population: One participant from the combined treatment-group was not included in the analysis due to withdrawal before the final collection of MDI-questionnaires.
Measure: Median (Inter-Quartile Range); unit: MDI-score
Arm/Group | Combined Treatment. | Denosumab Monotherapy | Placebo
Number analyzed (Participants) | 14 | 16 | 15
MDI-score | 0.0 [-4.0 to 1.0] | -0.5 [-4.5 to 1.0] | 0.0 [-3.0 to 0.0]
Statistical Analysis 1: Comparison: Combined Treatment. vs Denosumab Monotherapy vs Placebo; Test type: Superiority; p = 0.83, Kruskal-Wallis

18. Secondary Outcome: Adverse Reactions.
Description: All participants filled in questionnaires regarding symptoms related to the treatment.
  Results are reported in the Adverse Events section.
Time Frame: Monthly up to one year.
Reporting Status: Not Posted

19. Secondary Outcome: Bone Mineral Content
Description: Measured at baseline and after one year at the lumbar spine and distal 1/3 of the non-dominant antebrachii.
Time Frame: Baseline, one year
Population: Data were not collected
Arm/Group | Combined Treatment. | Denosumab Monotherapy | Placebo
Number analyzed (Participants) | 0 | 0 | 0

20. Secondary Outcome: Change in Cortical Width.
Description: Measured at baseline and after one year at the distal non-dominant antebrachii.
Time Frame: Baseline, one year.
Population: One participant from the combined treatment-group was not included in the analysis due to withdrawal before the final scan. One participant from the denosumab group experienced a wrist fracture prior to the final scan and was excluded. 4 patients did not provide data for the analysis due to errors in the technique of the obtained images.
Measure: Mean (Standard Error); unit: mm
Arm/Group | Combined Treatment. | Denosumab Monotherapy | Placebo
Number analyzed (Participants) | 12 | 14 | 14
mm | -0.04 (0.1) | 0.02 (0.08) | 0.04 (0.05)
Statistical Analysis 1: Comparison: Combined Treatment. vs Denosumab Monotherapy vs Placebo; Test type: Superiority; p > 0.05, ANOVA

21. Secondary Outcome: Change in Volumetric BMD for the Distal Forearm.
Description: Measured at baseline and after one year by QCT.
Time Frame: Baseline, one year
Population: One participant from the combined treatment-group was not included in the analysis due to withdrawal before the final scan. One participant from the denosumab group experienced a wrist fracture prior to the final scan and was excluded. 5 patients did not provide data for the analysis due to errors in the technique of the obtained images.
Measure: Mean (Standard Error); unit: mg/cm^3
Arm/Group | Combined Treatment. | Denosumab Monotherapy | Placebo
Number analyzed (Participants) | 12 | 13 | 14
mg/cm^3 | 1.0 (2.1) | 9.6 (3.7) | -1.1 (4.6)
Statistical Analysis 1: Comparison: Combined Treatment. vs Denosumab Monotherapy vs Placebo; Test type: Superiority; p = 0.0077, ANOVA

22. Secondary Outcome: Percentage Change in Volumetric BMD for the Lumbar Spine.
Description: Measured at baseline and after one year by QCT.
Time Frame: Baseline, one year
Population: as for outcome 9
Measure: Mean (Standard Error); unit: % change
Arm/Group | Combined Treatment. | Denosumab Monotherapy | Placebo
Number analyzed (Participants) | 13 | 16 | 15
% change | 6.18 (3.14) | 5.66 (1.85) | -2.94 (1.96)
Statistical Analysis 1: Comparison: Combined Treatment. vs Denosumab Monotherapy vs Placebo; Test type: Superiority; p = 0.011, ANOVA

23. Secondary Outcome: Percentage Change in Volumetric BMD for the Distal Forearm.
Description: Measured at baseline and after one year by QCT.
Time Frame: Baseline, one year
Population: as for outcome 21
Measure: Mean (Standard Error); unit: % change
Arm/Group | Combined Treatment. | Denosumab Monotherapy | Placebo
Number analyzed (Participants) | 12 | 13 | 14
% change | 0.53 (1.2) | 5.2 (1.0) | -0.74 (2.6)
Statistical Analysis 1: Comparison: Combined Treatment. vs Denosumab Monotherapy vs Placebo; Test type: Superiority; p = 0.011, ANOVA

24. Secondary Outcome: Mean p-PTH During Treatment.
Description: Blood samples were acquired once every 4 weeks for safety-purposes.
Time Frame: Monthly up to one year.
Measure: Median (95% Confidence Interval); unit: pmol/l
Units Other Than Participants: p-PTH measurements
Arm/Group | Combined Treatment. | Denosumab Monotherapy | Placebo
Number analyzed (Participants) | 15 | 16 | 15
Number analyzed (p-PTH measurements) | 211 | 240 | 225
pmol/l | 12.0 [11.1 to 12.9] | 13.4 [12.7 to 14.2] | 9.9 [9.5 to 10.4]
Statistical Analysis 1: Comparison: Combined Treatment. vs Denosumab Monotherapy vs Placebo; Test type: Superiority; p = 0.0001, Kruskal-Wallis

25. Secondary Outcome: Mean p-Phosphate During Treatment.
Description: Blood samples were acquired once every 4 weeks for safety-purposes.
Time Frame: Monthly up to one year.
Measure: Mean (Standard Error); unit: pmol/l
Units Other Than Participants: p-phosphate measurements
Arm/Group | Combined Treatment. | Denosumab Monotherapy | Placebo
Number analyzed (Participants) | 15 | 16 | 15
Number analyzed (p-phosphate measurements) | 211 | 240 | 225
pmol/l | 0.83 (0.013) | 0.76 (0.012) | 0.083 (0.011)
Statistical Analysis 1: Comparison: Combined Treatment. vs Denosumab Monotherapy vs Placebo; Test type: Superiority; p < 0.00001, ANOVA

26. Secondary Outcome: Percent Change From Baseline in p-N-terminal Propeptide of Type I Procollagen (p-P1NP).
Description: p-P1NP, change from baseline at 48 weeks.
Time Frame: Change from baseline at 48 weeks reported.
Population: as for outcome 11
Measure: Median (Inter-Quartile Range); unit: % change
Arm/Group | Combined Treatment. | Denosumab Monotherapy | Placebo
Number analyzed (Participants) | 14 | 16 | 15
% change | -63.1 [-66.9 to -57.2] | -66.1 [-75.9 to -55.4] | 17.8 [-11.0 to 31.5]
Statistical Analysis 1: Comparison: Combined Treatment. vs Denosumab Monotherapy vs Placebo; Test type: Superiority; p = 0.0001, Kruskal-Wallis

27. Secondary Outcome: Percent Change From Baseline in P-osteocalcin.
Description: p-osteocalcin, change from baseline at 48 weeks.
Time Frame: Change from baseline at 48 weeks reported.
Population: as for outcome 11
Measure: Median (Inter-Quartile Range); unit: % change
Arm/Group | Combined Treatment. | Denosumab Monotherapy | Placebo
Number analyzed (Participants) | 14 | 16 | 15
% change | -60.0 [-69.8 to -36.9] | -58.9 [-66.9 to -49.0] | 7.0 [-0.9 to 36.9]
Statistical Analysis 1: Comparison: Combined Treatment. vs Denosumab Monotherapy vs Placebo; Test type: Superiority; p = 0.0001, ANOVA

28. Secondary Outcome: Percent Change From Baseline in S-bone-specific Alkaline Phosphatase (BAP).
Description: S-Bone specific alkaline phosphatase, change from baseline at 48 weeks.
Time Frame: Change from baseline at 48 weeks reported.
Population: as for outcome 11
Measure: Median (Inter-Quartile Range); unit: % change
Arm/Group | Combined Treatment. | Denosumab Monotherapy | Placebo
Number analyzed (Participants) | 14 | 16 | 15
% change | -40.0 [-46.3 to -24.1] | -46.3 [-51.5 to -38.4] | 9.7 [-7.9 to 32.5]
Statistical Analysis 1: Comparison: Combined Treatment. vs Denosumab Monotherapy vs Placebo; Test type: Superiority; p = 0.0001, Kruskal-Wallis

29. Secondary Outcome: Percent Change From Baseline in p-Tartrate-resistant Acid Phosphatase 5b (Trap5b).
Description: P-Trap5b, change from baseline at 48 weeks.
Time Frame: Change from baseline at 48 weeks reported.
Population: as for outcome 11
Measure: Median (Inter-Quartile Range); unit: % change
Arm/Group | Combined Treatment. | Denosumab Monotherapy | Placebo
Number analyzed (Participants) | 14 | 16 | 15
% change | -27.8 [-34.1 to -2.3] | -36.7 [-51.8 to -16.4] | 2.3 [-4.9 to 19.6]

30. Secondary Outcome: Percent Change From Baseline in p-Sclerostin.
Description: P-Sclerostin, change from baseline at 48 weeks.
Time Frame: Change from baseline at 48 weeks reported.
Population: as for outcome 11
Measure: Median (Inter-Quartile Range); unit: % change
Arm/Group | Combined Treatment. | Denosumab Monotherapy | Placebo
Number analyzed (Participants) | 14 | 16 | 15
% change | 10.0 [3.1 to 21.1] | 6.5 [0.9 to 15.9] | 4.8 [-2.3 to 13.9]
Statistical Analysis 1: Comparison: Combined Treatment. vs Denosumab Monotherapy vs Placebo; Test type: Superiority; p = 0.5, Kruskal-Wallis

31. Secondary Outcome: Percent Change From Baseline in P-fibroblast Growth Factor 23 (FGF23).
Description: P-FGF23 , change from baseline at 48 weeks.
Time Frame: Change from baseline at 48 weeks reported.
Population: as for outcome 11
Measure: Median (Inter-Quartile Range); unit: % change
Arm/Group | Combined Treatment. | Denosumab Monotherapy | Placebo
Number analyzed (Participants) | 14 | 16 | 15
% change | 35.8 [0.0 to 52.9] | 20.4 [-13.6 to 58.2] | 28.0 [-25.9 to 64.7]
Statistical Analysis 1: Comparison: Combined Treatment. vs Denosumab Monotherapy vs Placebo; Test type: Superiority; p = 0.85, ANOVA

32. Secondary Outcome: Changes in p-25-vitamin D
Description: P-25-vitD , change from baseline at 48 weeks.
Time Frame: Change from baseline at 48 weeks reported.
Population: as for outcome 11
Measure: Median (Inter-Quartile Range); unit: nmol/l
Arm/Group | Combined Treatment. | Denosumab Monotherapy | Placebo
Number analyzed (Participants) | 14 | 16 | 15
nmol/l | 22.1 [13.3 to 32.6] | 16.0 [4.1 to 22.0] | 21.2 [8.2 to 30.5]
Statistical Analysis 1: Comparison: Combined Treatment. vs Denosumab Monotherapy vs Placebo; Test type: Superiority; p = 0.22, ANOVA

33. Secondary Outcome: Changes in s-1,25-vitamin D
Description: S-1,25-vitD, change from baseline at 48 weeks.
Time Frame: Change from baseline at 48 weeks reported.
Population: as for outcome 11
Measure: Median (Inter-Quartile Range); unit: pmol/l
Arm/Group | Combined Treatment. | Denosumab Monotherapy | Placebo
Number analyzed (Participants) | 14 | 16 | 15
pmol/l | 7.5 [-4.0 to 35.0] | 4.5 [-15.0 to 25.5] | 26.0 [14.0 to 36.0]
Statistical Analysis 1: Comparison: Combined Treatment. vs Denosumab Monotherapy vs Placebo; Test type: Superiority; p = 0.18, Kruskal-Wallis

34. Secondary Outcome: Patients With Nephrocalcinosis, Final Scan.
Description: Number of subjects w. renal calcifications at final scan.
Time Frame: Baseline, one year
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Combined Treatment. | Denosumab Monotherapy | Placebo
Number analyzed (Participants) | 14 | 16 | 15
Participants | 2 | 1 | 3

35. Other Pre Specified Outcome: Safety Measures
Description: Biochemical measures of changes in liver, infection, kidney and electrolyte-status and urinary excretion of calcium.
Time Frame: Monthly up to one year.
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events were collected for each participant from baseline until two weeks after treatment-cessation, up to 1 year.
Description: Adverse events were collected at each visit using a adverse event questionnaire as well as assessment by a study-physician.
Arm/Group | Combined Treatment. | Denosumab Monotherapy | Placebo
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/16 | 0/15
Serious Adverse Events (participants affected / at risk) | 2/15 | 1/16 | 3/15
Other Adverse Events (participants affected / at risk) | 13/15 | 15/16 | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Combined Treatment. (N=15) | Denosumab Monotherapy (N=16) | Placebo (N=15)
Angina, Unstable (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Polycythaemia Vera (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Epilepsy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Inflammatory Bowel Disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Erysipelas (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Combined Treatment. (N=15) | Denosumab Monotherapy (N=16) | Placebo (N=15)
Leg edema (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (7) | 0 (0)
Coughing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (9) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (6) | 0 (0)
Paraesthesia, hands (Nervous system disorders) | 6 (36) | 3 (15) | 4 (20)
Paraesthesia, feet (Nervous system disorders) | 4 (17) | 3 (27) | 2 (23)
Headache (Nervous system disorders) | 2 (4) | 1 (1) | 1 (1)
Fatigue (General disorders) | 1 (2) | 1 (2) | 2 (5)
Dizziness (Ear and labyrinth disorders) | 1 (3) | 4 (7) | 3 (17)
Nausea (Gastrointestinal disorders) | 7 (18) | 9 (21) | 4 (5)
Abdominal pain (Gastrointestinal disorders) | 2 (6) | 2 (6) | 1 (1)
Gastroenteritis (Gastrointestinal disorders) | 3 (5) | 0 (0) | 2 (2)
Cystitis (Renal and urinary disorders) | 2 (2) | 1 (5) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 6 (14) | 6 (17) | 3 (20)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (12) | 1 (1) | 1 (1)
Hypocalcaemia (Endocrine disorders) | 6 (33) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 5 (12) | 6 (20) | 4 (5)

LIMITATIONS AND CAVEATS:
Important limitations are the relatively small number of study-participants, and the lack of a cinacalcet monotherapy-arm.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-10): https://cdn.clinicaltrials.gov/large-docs/57/NCT03027557/Prot_SAP_000.pdf